CLINICAL TRIAL: NCT00366210
Title: Constraint-Induced Therapy Modified for Rehabilitating Arm Function in Stroke Survivors w/Plegic Hands
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F060112013
Record Dates: First submitted 2006-08-18; First posted 2006-08-21 (Estimated); Last update posted 2014-12-25 (Estimated); Status verified 2010-08

CONDITIONS: Chronic Stroke Survivors With Plegic Hand
Keywords: stroke; rehabilitation; physical therapy; occupational therapy; arm
MeSH Terms: conditions — Stroke | interventions — Therapeutics; Biofeedback, Psychology

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Expanded CI therapy (Experimental): 3.5 hours of training for the more-affected arm set in the laboratory for 15 consecutive weekdays
  Interventions: Behavioral: Constraint-Induced Movement (CI) Therapy
- Placebo Control (Placebo Comparator): Stretching, movement exercises, and EMG biofeedback for the same duration as the experimental intervention.
  Interventions: Behavioral: Stretching, Relaxation, & Biofeedback
- Usual & Customary Care Control (No Intervention): Treatments available to participants as part of their regular medical care, such as conventional physical or occupational therapy. For some participants, this would involve no treatment, since all participants were more than one year post stroke.f standard clinical care.

INTERVENTIONS:
Behavioral: Constraint-Induced Movement (CI) Therapy
  Arms: Expanded CI therapy
Behavioral: Stretching, Relaxation, & Biofeedback — Passive stretching of both arms, EMG biofeedback for more-impaired arm
  Arms: Placebo Control

SUMMARY:
The purpose of this study is to compare modified CI therapy for strokes survivors with very limited function to an alternative package of conventional physical rehabilitation techniques

DETAILED DESCRIPTION:
Constraint-Induced Movement therapy or CI therapy is a rehabilitation method, based on behavioral neuroscience studies of deafferented monkeys, that has been shown in controlled studies to produce large improvements in real-world upper-extremity use in individuals with chronic stroke. Up till now, survivors of stroke with plegic hands have been excluded from CI therapy protocols, whether on a research or clinical basis. Such individuals are estimated to make up at least 35% of the population with chronic stroke with residual motor deficit. Furthermore, there are no other interventions for such individuals that have controlled evidence of efficacy for increasing real-world function. Thus, these stroke survivors represent a large number of healthcare consumers with limited treatment options.

We recently completed a pilot study of a modified form of CI therapy for stroke survivors with plegic hands, and obtained surprisingly positive findings. Six individuals were enrolled who had a flicker of active movement at the elbow and at the wrist or a finger and 30° of active range of motion at the shoulder. Participants received three weeks of CI therapy, combined with other modes of therapy, for six hours per day. The treatment package included tone management/movement facilitation, training of more-impaired arm use using shaping, functional task practice, restraint of the less-impaired arm in the laboratory and at home as indicated, and a package of behavioral methods for transferring gains from the laboratory to the home situation. As a group, the patients showed a large improvement in more-impaired arm use in daily life after treatment (Motor Activity Log or MAL; p's < 05, Effect Size > 1.5). Improvements in more-impaired arm motor ability, as measured by scores on a laboratory motor performance test (graded Wolf Motor Function Test; gWMFT) and standardized clinical examination (Fugl-Meyer), were also substantial (p's < .05).

Based on these initial findings, we propose a randomized, controlled clinical trial to rigorously test the efficacy of this modification of CI therapy for rehabilitating arm function in chronic stroke patients with severe upper-extremity impairment. To this end, 40 survivors of stroke with plegic hands will be randomly assigned to receive the intervention described above or a placebo control procedure of the same duration. Control participants will receive either 1) tone management, EMG biofeedback and other procedures in alternating blocks for 6 hr daily for 15 consecutive weekdays or 2) usual & customary care. Measures of arm motor ability (gWMFT; Fugl-Meyer), arm use in daily life (MAL, accelerometry), and quality of life (Stroke Impact Scale) will be administered to all participants before and after treatment and at long-term. If the modified CI therapy participants shows larger improvements in more-impaired arm function than the control group participants, this will suggest it is an efficacious treatment and raise hopes of additional recovery for a large group of healthcare consumers with limited treatment options.

ELIGIBILITY:
Inclusion Criteria:

1a. The ability to initiate extension against gravity at the wrist or at least one digit and initiate extension and flexion at the elbow.

1b. No active movement required for the wrist, fingers or thumb. At least 20° active extension required at elbow.

2. Actively move the shoulder at least 30 degrees in flexion, abduction, or scaption 3. Score less than 4 on the Modified Ashworth Scale for all impaired joints 4. Passive range of motion criteria > or equal to 90° shoulder flexion, > or equal to 90° shoulder abduction, > or equal to 45° shoulder external rotation, < or equal to 30° short of normal elbow extension, forearm supination to at least neutral, forearm pronation 45° or more from neutral, < equal to 35° short of normal wrist extension, and < equal to 35° short of normal metacarpophalangeal extension on all the digits.

Other Exclusion Criteria. Among the principal exclusion criteria are:

1. Less than 6 months post-stroke.
2. Motor problems that are not primarily unilateral.
3. Other neurological or musculoskeletal conditions, including excessive pain, affecting UE function.
4. Insufficient stamina or serious uncontrolled medical problems.
5. Serious cognitive deficits including inadequate ability to follow test instructions.
6. Less than 19 years old. Grade 4 MMC for wrist, thumb, fingers; i.e., individuals who can actively extend the wrist > or equal to 10°, abduct the thumb or equal to 10°, and initiate extension of at least two additional digits will be excluded.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2005-10; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Motor Activity Log | Pre-treatment, Post-treatment, followup

CONTACTS AND LOCATIONS:
Overall Officials: Gitendra Uswatte, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States